CLINICAL TRIAL: NCT00734656
Title: Subjective and Physiological Effects of Alcohol: Role of Genetic Variation and Adrenal Hormones
Brief Title: Pharmacogenetics of Alcohol: Treatment Implications
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UConn Health (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Jonathan Covault, Associate Professor, UConn Health
Allocation: Randomized | Model: Factorial | Masking: Quadruple
Other Study IDs: 06-218S-2; 619 (Other Grant/Funding Number: GCRC); 5R01AA015606-02 (NIH)
Record Dates: First submitted 2008-07-31; First posted 2008-08-14 (Estimated); Results first posted 2012-03-27 (Estimated); Last update posted 2012-03-28 (Estimated); Status verified 2012-03

CONDITIONS: Alcohol Related Disorders; Alcoholism; Alcohol Abuse
Keywords: steroid 5Alpha Reductase; dutasteride; neuroactive steroid
MeSH Terms: conditions — Alcohol-Related Disorders; Alcoholism | interventions — Dutasteride; Ethanol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Placebo medication + placebo alcohol (Placebo Comparator)
  Interventions: Drug: placebo medication + placebo alcohol
- Placebo Medication + 0.8 gr/kg Ethanol (Experimental)
  Interventions: Drug: placebo medication + ethanol
- 4 mg Dutasteride + Placebo Alcohol (Experimental)
  Interventions: Drug: dutasteride + placebo alcohol
- 4 mg Dutasteride + 0.8 gr/kg Ethanol (Experimental)
  Interventions: Drug: dutasteride + ethanol

INTERVENTIONS:
Drug: dutasteride + ethanol — 4 mg dutasteride administered 2-4 days prior to ingestion of 0.8 mg/kg ethanol divided between three drinks consumed over 36 minutes
  Other Names: Avodart
  Arms: 4 mg Dutasteride + 0.8 gr/kg Ethanol
Drug: placebo medication + ethanol — placebo medication administered 2-4 days prior to ingestion of 0.8 gr/kg ethanol divided between three drinks consumed over 36 minutes
  Arms: Placebo Medication + 0.8 gr/kg Ethanol
Drug: dutasteride + placebo alcohol — 4 mg dutasteride administered 2-4 days prior to ingestion of three drinks each containing 1 cc ethanol consumed over 36 minutes
  Other Names: Avodart
  Arms: 4 mg Dutasteride + Placebo Alcohol
Drug: placebo medication + placebo alcohol — placebo medication administered 2-4 days prior to ingestion of three drinks each containing 1 cc ethanol consumed over 36 minutes
  Arms: Placebo medication + placebo alcohol

SUMMARY:
This study will explore the hypothesis that effects of alcohol are in part mediated by increased production of neuroactive steroids, which interact with GABAA-receptors. We propose to study non-dependent drinkers using a 4-session within-subjects design in which alcohol / placebo is paired with dutasteride / placebo pretreatment. Dutasteride is a 5-alpha steroid reductase (5AR) inhibitor that limits the production of dihydrotestosterone and the 5a-reduced neuroactive steroids allopregnanolone, pregnanolone and 3a,5a-androstanediol.

DETAILED DESCRIPTION:
Alcohol has multiple pharmacological effects, though which of these effects relate to the risk of alcohol dependence is not clear. Animal studies indicate that the neuroactive steroid allopregnanolone is an alcohol-modulated endogenous agonist at GABAA receptors and that genetic variation in steroid 5a-reductase type I gene which generates neuroactive steroids, may moderate alcohol effects. To better define the role of neuroactive steroids we will conduct a laboratory study of non-alcohol dependent drinkers using a 4-session design in which alcohol/placebo beverage is paired with dutasteride/placebo pretreatment. Dutasteride, an inhibitor of both type I and type II 5a-reductase enzymes, blocks the production of 5a-reduced neuroactive steroids. This study will extend our preliminary findings with finasteride by including a) a placebo control for alcohol, b) a more specific inhibitor of both 5a-reductase isoenzymes, c) a larger group of subjects (including both light and heavy drinkers).

ELIGIBILITY:
Inclusion Criteria:

* Main Study: Subjects will be healthy volunteers with or without parental history of alcoholism who are 21-45 years old and who have a BMI >18.5 and <32.5. Drinking history: All subjects must report at least one occasion in the prior month of drinking at least 3 drinks on a single day; additionally, LD subjects will be selected if they drink 1-3 drinks, 1-3 times per week (up to 5 drinks per week on average), with no more than one occasion in the past 2 months on which they drank >4 drinks. HD subjects will be selected if they report drinking at least 10 drinks per week, with at least one episode per week of heavy drinking.

Exclusion Criteria:

* Main Study: Subjects cannot have a current or past DSM-IV diagnosis of alcohol or drug dependence, current or past 24-months diagnosis of alcohol or drug abuse or another major psychiatric disorder, neurological illness, have had a hypersensitivity reaction to dutasteride, evidence of liver dysfunction, currently be using benzodiazepines, other psychotropic medications or medications that are known to influence steroid hormone levels or metabolism or modify the effects of alcohol. Nicotine-dependent subjects will be excluded to avoid the confounding effects of nicotine withdrawal during day-long laboratory sessions. Women are not allowed to participate. Subjects anticipating moving from the area during the period of their planned study participation will be excluded from study entry.

Ages: 21 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 94 (Actual)
Dates: Start 2007-03; Primary Completion 2010-10 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Covault, MD, PhD, Principal Investigator — UConn Health
Locations (1):
- University of Connecticut Health Center, Farmington, Connecticut, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Non-treatment seeking social drinkers recruited from community settings 2007-2010.
Pre-assignment Details: A total of 148 subjects enrolled, 31 subjects were excluded for not meeting entrance criteria, 23 subjects withdrew before first dose of study medication. 94 subjects were randomized to one of 24 possible laboratory session sequences for exposure to each of 4 treatment conditions.
Groups:
- Placebo Medication + Placebo Alcohol: placebo medication paired with placebo alcohol
- Placebo Medication + 0.8 gr/kg Ethanol: placebo medication paired with active alcohol
- 4 mg Dutasteride + Placebo Alcohol: 4 mg dutasteride paired with placebo alcohol
- 4 mg Dutasteride + 0.8 mg/kg Ethanol: 4 mg dutasteride paired with active alcohol
Period: Lab Session 1
Arm/Group | Placebo Medication + Placebo Alcohol | Placebo Medication + 0.8 gr/kg Ethanol | 4 mg Dutasteride + Placebo Alcohol | 4 mg Dutasteride + 0.8 mg/kg Ethanol
Started | 24 | 23 | 26 | 21
Completed | 22 | 23 | 26 | 21
Not Completed | 2 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 0 | 0 | 0
Period: Washout 1
Arm/Group | Placebo Medication + Placebo Alcohol | Placebo Medication + 0.8 gr/kg Ethanol | 4 mg Dutasteride + Placebo Alcohol | 4 mg Dutasteride + 0.8 mg/kg Ethanol
Started | 22 | 23 | 26 | 21
Completed | 21 | 18 | 24 | 18
Not Completed | 1 | 5 | 2 | 3
Not completed — Withdrawal by Subject | 1 | 5 | 2 | 3
Period: Lab Session 2
Arm/Group | Placebo Medication + Placebo Alcohol | Placebo Medication + 0.8 gr/kg Ethanol | 4 mg Dutasteride + Placebo Alcohol | 4 mg Dutasteride + 0.8 mg/kg Ethanol
Started | 19 (subjects cross-over to different treatment condition with each lab session in factorial design,) | 21 (subjects cross-over to different treatment condition with each lab session in factorial design,) | 21 (subjects cross-over to different treatment condition with each lab session in factorial design,) | 20 (subjects cross-over to different treatment condition with each lab session in factorial design,)
Completed | 18 | 21 | 21 | 19
Not Completed | 1 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 1
Period: Washout 2
Arm/Group | Placebo Medication + Placebo Alcohol | Placebo Medication + 0.8 gr/kg Ethanol | 4 mg Dutasteride + Placebo Alcohol | 4 mg Dutasteride + 0.8 mg/kg Ethanol
Started | 18 | 21 | 21 | 19
Completed | 17 | 20 | 20 | 19
Not Completed | 1 | 1 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 1 | 0
Period: Lab Session 3
Arm/Group | Placebo Medication + Placebo Alcohol | Placebo Medication + 0.8 gr/kg Ethanol | 4 mg Dutasteride + Placebo Alcohol | 4 mg Dutasteride + 0.8 mg/kg Ethanol
Started | 18 (subjects cross-over to different treatment condition with each lab session in factorial design,) | 19 (subjects cross-over to different treatment condition with each lab session in factorial design,) | 20 (subjects cross-over to different treatment condition with each lab session in factorial design,) | 19 (subjects cross-over to different treatment condition with each lab session in factorial design,)
Completed | 18 | 19 | 20 | 19
Not Completed | 0 | 0 | 0 | 0
Period: Washout 3
Arm/Group | Placebo Medication + Placebo Alcohol | Placebo Medication + 0.8 gr/kg Ethanol | 4 mg Dutasteride + Placebo Alcohol | 4 mg Dutasteride + 0.8 mg/kg Ethanol
Started | 18 | 19 | 20 | 19
Completed | 17 | 19 | 20 | 18
Not Completed | 1 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 1
Period: Lab Session 4
Arm/Group | Placebo Medication + Placebo Alcohol | Placebo Medication + 0.8 gr/kg Ethanol | 4 mg Dutasteride + Placebo Alcohol | 4 mg Dutasteride + 0.8 mg/kg Ethanol
Started | 20 (subjects cross-over to different treatment condition with each lab session in factorial design,) | 18 (subjects cross-over to different treatment condition with each lab session in factorial design,) | 16 (subjects cross-over to different treatment condition with each lab session in factorial design,) | 20 (subjects cross-over to different treatment condition with each lab session in factorial design,)
Completed | 20 | 18 | 16 | 19
Not Completed | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: All study participants enrolled in Lab Session 1
Arm/Group | All Study Participants
Number analyzed (Participants) | 94
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 94
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 26.1 (6.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 94
Region of Enrollment [Number; unit: participants]
  United States | 94

OUTCOME MEASURES:

1. Primary Outcome: Breath Alcohol
Description: Breath Alcohol level
Time Frame: 40 minutes after beginning drink
Population: Subjects who completed all 4 arms of study (e.g. completed each combination of dutasteride or placebo paired with 0.8 gr/kg ethanol or alcohol flavor mask)less 3 subjects removed during data cleaning due to pharmacy errors (n=2) or protocol deviation (n=1)resulted in 70 subjects completing each condition for analysis.
Measure: Mean (Standard Error); unit: gr/dL
Arm/Group | Placebo Medication + Placebo Alcohol | Placebo Medication + 0.8 gr/kg Ethanol | 4 mg Dutasteride + Placebo Alcohol | 4 mg Dutasteride + 0.8 mg/kg Ethanol
Number analyzed (Participants) | 70 | 70 | 70 | 70
gr/dL | 0.001 (0.0004) | 0.075 (0.003) | 0.001 (0.0005) | 0.071 (0.003)
Statistical Analysis 1: Comparison: Placebo Medication + 0.8 gr/kg Ethanol vs 4 mg Dutasteride + 0.8 mg/kg Ethanol; null hypothesis - dutasteride does not affect blood alcohol following standardized dose of alcohol (0.8 gr/kg); Test type: Superiority or Other; p = 0.28, t-test, 2 sided

2. Primary Outcome: BAES Sedation Response, Average of 6 Time Points
Description: Biphasic Alcohol Effects Scale (BAES) Sedation items - sum of subjective responses - 0(not at all)to 10 (extremely)- for 7 sedation related questions regarding effects of alcohol. Total BAES sedation subscale score 0-70 with higher numbers indicating greater sedative effects of alcohol. [Martin, C. S., M. Earleywine, R. E. Musty, M. W. Perrine and R. M. Swift (1993a). Development and validation of the Biphasic Alcohol Effects Scale. Alcohol Clin Exp Res 17(1): 140-6.]
Time Frame: 40, 80, 120, 160, 210 and 240 minutes after start of drinking
Population: as for outcome 1
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo Medication + Placebo Alcohol | Placebo Medication + 0.8 gr/kg Ethanol | 4 mg Dutasteride + Placebo Alcohol | 4 mg Dutasteride + 0.8 mg/kg Ethanol
Number analyzed (Participants) | 70 | 70 | 70 | 70
units on a scale | 0.7 (0.1) | 8.9 (0.6) | 1.5 (0.2) | 7.4 (0.5)
Statistical Analysis 1: Comparison: Placebo Medication + 0.8 gr/kg Ethanol vs 4 mg Dutasteride + 0.8 mg/kg Ethanol; null hypothesis: dutasteride pre-treatment does not reduce the sedative effect of alcohol; Test type: Superiority or Other; p = 0.010, Mixed Models Analysis

3. Primary Outcome: BAES Stimulation Response, Average of 6 Time Points
Description: Biphasic Alcohol Effects Scale (BAES)Simulation items - sum of subjective responses - 0(not at all)to 10 (extremely)- for 7 stimulation related questions regarding effects of alcohol. Total BAES stimulation subscale score 0-70 with higher numbers indicating greater stimulating effects of alcohol. [Martin, C. S., M. Earleywine, R. E. Musty, M. W. Perrine and R. M. Swift (1993a). Development and validation of the Biphasic Alcohol Effects Scale. Alcohol Clin Exp Res 17(1): 140-6.]
Time Frame: 40, 80, 120, 160, 210 and 240 minutes after start of drinking
Population: as for outcome 1
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo Medication + Placebo Alcohol | Placebo Medication + 0.8 gr/kg Ethanol | 4 mg Dutasteride + Placebo Alcohol | 4 mg Dutasteride + 0.8 mg/kg Ethanol
Number analyzed (Participants) | 70 | 70 | 70 | 70
units on a scale | 0.7 (0.1) | 4.2 (0.4) | 1.7 (0.3) | 4.8 (0.4)
Statistical Analysis 1: Comparison: Placebo Medication + 0.8 gr/kg Ethanol vs 4 mg Dutasteride + 0.8 mg/kg Ethanol; null hypothesis: dutasteride pre-treatment does not reduce the stimulating effect of alcohol; Test type: Superiority or Other; p = 0.17, Mixed Models Analysis

4. Secondary Outcome: Change in Serum 3a-androstanediol Glucuronide
Description: Ratio of serum 3a-androstanediol drawn prior to alcohol administration (2-4 days after medication administration) compared to the baseline level prior to medication dose. The pharmacologic effect of dutasteride was measured by assay of serum 5a-androstan-3a,17b-diol,17-glucuronide (aka 3a-androstanediol glucuronide) as a biochemical measure of 5a-reductase enzyme inhibition. 3a-androstanediol glucuronide is the primary metabolic excretion product of 3a,5a-androstane neuroactive steroids. The
Time Frame: Baseline (pre medication administration) and 2-4 days post-medication (alcohol session)
Population: as for outcome 1
Measure: Mean (Standard Error); unit: ratio
Arm/Group | Placebo Medication + Placebo Alcohol | Placebo Medication + 0.8 gr/kg Ethanol | 4 mg Dutasteride + Placebo Alcohol | 4 mg Dutasteride + 0.8 mg/kg Ethanol
Number analyzed (Participants) | 70 | 70 | 70 | 70
ratio | 1.04 (0.033) | 1.11 (0.03) | 0.31 (0.02) | 0.31 (0.02)
Statistical Analysis 1: Comparison: Placebo Medication + 0.8 gr/kg Ethanol vs 4 mg Dutasteride + 0.8 mg/kg Ethanol; null hypothesis - A single 4 mg dose of dutasteride does not reduce serum 3a-androstanediol glucuronide levels; Test type: Superiority or Other; p < 0.001, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 2-11 days following medication administration. In person at time of alcohol laboratory session (2-4 days after medication dose)and by phone 1-day and 1-week following alcohol laboratory session.
Arm/Group | Placebo Medication + Placebo Alcohol | Placebo Medication + 0.8 gr/kg Ethanol | 4 mg Dutasteride + Placebo Alcohol | 4 mg Dutasteride + 0.8 mg/kg Ethanol
Serious Adverse Events (participants affected / at risk) | 0/78 | 0/81 | 0/83 | 0/78
Other Adverse Events (participants affected / at risk) | 9/78 | 8/81 | 11/83 | 12/78
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Medication + Placebo Alcohol (N=78) | Placebo Medication + 0.8 gr/kg Ethanol (N=81) | 4 mg Dutasteride + Placebo Alcohol (N=83) | 4 mg Dutasteride + 0.8 mg/kg Ethanol (N=78)
Fatigue (General disorders) | 2 (2) | 2 (2) | 2 (3) | 1 (1)
Headace (Nervous system disorders) | 2 (2) | 3 (3) | 1 (1) | 3 (3)
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2) | 2 (2)
Libido, reduced (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Stomach discomfort (Gastrointestinal disorders) | 2 (2) | 2 (2) | 4 (5) | 6 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes